CLINICAL TRIAL: NCT02493504
Title: Effects of Heparin on Early Patency of Arteriovenous Fistula in Angioaccess Surgery of Patients With End-Stage Renal Disease
Brief Title: Effects of Heparin on Arteriovenous Fistula Patency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fatemeh Hoseinzadegan (Other)
Responsible Party: Sponsor-Investigator, Fatemeh Hoseinzadegan, Dr., Shahid Beheshti University of Medical Sciences
Organization: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHBMU-001124
Record Dates: First submitted 2015-07-01; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Arteriovenous Fistula
Keywords: Heparin
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heparin (Experimental): 75 patients were randomly assigned to receive 100units/kg of heparin after dissection prior to anastomosis.
  Interventions: Drug: Heparin
- Control (No Intervention): 75 received no intraoperative heparin injection.

INTERVENTIONS:
Drug: Heparin — 100units/kg of heparin were administered for the case group after dissection prior to anastomosis.
  Other Names: Case
  Arms: Heparin

SUMMARY:
Arteriovenous fistula (AVF) is now the optimal method of obtaining vascular access for dialysis. Measures such as systemic anticoagulation have been proposed as means of increasing patency rates but enough evidence does not exist to support their use. The investigators aimed to evaluate the efficacy of preoperative heparin injection on patency of AVF during the first 24 hours after surgery and to determine whether such measure can be used to prevent early thrombosis of the vascular access.

DETAILED DESCRIPTION:
The study was carried out on patients admitted to Shohada-e-Tajrish hospital for permanent vascular access placement since April 2011 through September 2012. The exclusion criteria consisted of having a contraindication of administration of anticuagulant agent. 150 patients were enrolled in the study.

All patients were operated on by a single surgeon (Dr Mozafar. The non dominant upper extremity (mostly the left arm) was generally used unless unfavorable vasculature or previous fistula placement changed the preference. The anastomosis technique was either end-to-side or side-to-side using a number 6.0 prolene suture. 75 patients were randomly assigned to receive 100units/kg of heparin after dissection prior to anastomosis while the other 75 received no intraoperative heparin injection. Auscultation of bruit and palpation of thrill was used to assess arteriovenous fistula patency in the first 24 hours after AVF placement.

Data analysis was performed using SPSS v.20. A p-value of less than 0.05 was considered as statistically significant. Bivariate analysis in the form of Chi-square tests, T-test and Fischer's exact test were calculated.

Patient enrollment was voluntary and no costs were imposed on the patients. The study protocol was in accordance with 1975 Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease, In need of AVF placement

Exclusion Criteria:

* Contraindications for anticoagulant therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The number of patients with a bruit auscultated over AVF | The first 24 hours after anostomosis
  Hearing a bruit through auscultation over the AVF is regarded as a positive measure or in other words a patent AVF. The frequency of positive measures are compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Mozafar, M.D., Study Director — Associate Professor of General and Vascular Surgery

REFERENCES:
- [Background] Zhang QL, Rothenbacher D. Prevalence of chronic kidney disease in population-based studies: systematic review. BMC Public Health. 2008 Apr 11;8:117. doi: 10.1186/1471-2458-8-117. PMID 18405348
- [Background] Allon M, Robbin ML. Increasing arteriovenous fistulas in hemodialysis patients: problems and solutions. Kidney Int. 2002 Oct;62(4):1109-24. doi: 10.1111/j.1523-1755.2002.kid551.x. PMID 12234281
- [Background] Haimov M, Baez A, Neff M, Slifkin R. Complications of arteriovenous fistulas for hemodialysis. Arch Surg. 1975 Jun;110(6):708-12. doi: 10.1001/archsurg.1975.01360120026004. No abstract available. PMID 1147768
- [Background] Perera GB, Mueller MP, Kubaska SM, Wilson SE, Lawrence PF, Fujitani RM. Superiority of autogenous arteriovenous hemodialysis access: maintenance of function with fewer secondary interventions. Ann Vasc Surg. 2004 Jan;18(1):66-73. doi: 10.1007/s10016-003-0094-y. Epub 2004 Jan 20. PMID 14727162
- [Background] Abularrage CJ, Sidawy AN, Weiswasser JM, White PW, Arora S. Medical factors affecting patency of arteriovenous access. Semin Vasc Surg. 2004 Mar;17(1):25-31. doi: 10.1053/j.semvascsurg.2003.11.006. PMID 15011176
- [Background] Green LD, Lee DS, Kucey DS. A metaanalysis comparing surgical thrombectomy, mechanical thrombectomy, and pharmacomechanical thrombolysis for thrombosed dialysis grafts. J Vasc Surg. 2002 Nov;36(5):939-45. doi: 10.1067/mva.2002.127524. PMID 12422093
- [Background] Smith GE, Gohil R, Chetter IC. Factors affecting the patency of arteriovenous fistulas for dialysis access. J Vasc Surg. 2012 Mar;55(3):849-55. doi: 10.1016/j.jvs.2011.07.095. Epub 2011 Nov 8. PMID 22070937
- [Background] Erkut B, Unlu Y, Ceviz M, Becit N, Ates A, Colak A, Kocak H. Primary arteriovenous fistulas in the forearm for hemodialysis: effect of miscellaneous factors in fistula patency. Ren Fail. 2006;28(4):275-81. doi: 10.1080/08860220600583617. PMID 16771241
- [Background] Dember LM, Beck GJ, Allon M, Delmez JA, Dixon BS, Greenberg A, Himmelfarb J, Vazquez MA, Gassman JJ, Greene T, Radeva MK, Braden GL, Ikizler TA, Rocco MV, Davidson IJ, Kaufman JS, Meyers CM, Kusek JW, Feldman HI; Dialysis Access Consortium Study Group. Effect of clopidogrel on early failure of arteriovenous fistulas for hemodialysis: a randomized controlled trial. JAMA. 2008 May 14;299(18):2164-71. doi: 10.1001/jama.299.18.2164. PMID 18477783
- [Background] Ghorbani A, Aalamshah M, Shahbazian H, Ehsanpour A, Aref A. Randomized controlled trial of clopidogrel to prevent primary arteriovenous fistula failure in hemodialysis patients. Indian J Nephrol. 2009 Apr;19(2):57-61. doi: 10.4103/0971-4065.53323. PMID 20368925
- [Background] Akin EB, Topcu O, Ozcan H, Ersoz S, Aytac S, Anadol E. Hemodynamic effect of transdermal glyceryl trinitrate on newly constructed arteriovenous fistula. World J Surg. 2002 Oct;26(10):1256-9. doi: 10.1007/s00268-002-6515-1. Epub 2002 Sep 4. PMID 12205547
- [Background] Tessitore N, Bedogna V, Poli A, Mantovani W, Lipari G, Baggio E, Mansueto G, Lupo A. Adding access blood flow surveillance to clinical monitoring reduces thrombosis rates and costs, and improves fistula patency in the short term: a controlled cohort study. Nephrol Dial Transplant. 2008 Nov;23(11):3578-84. doi: 10.1093/ndt/gfn275. Epub 2008 May 29. PMID 18511608
- [Background] Sharathkumar A, Hirschl R, Pipe S, Crandell C, Adams B, Lin JJ. Primary thromboprophylaxis with heparins for arteriovenous fistula failure in pediatric patients. J Vasc Access. 2007 Oct-Dec;8(4):235-44. PMID 18161668
- [Background] Bhomi KK, Shrestha S, Bhattachan CL. Role of systemic anticoagulation in patients undergoing vascular access surgery. Nepal Med Coll J. 2008 Dec;10(4):222-4. PMID 19558057
- [Background] D'Ayala M, Smith RM, Martone C, Briggs W, Deitch JS, Wise L. The effect of systemic anticoagulation in patients undergoing angioaccess surgery. Ann Vasc Surg. 2008 Jan;22(1):11-5. doi: 10.1016/j.avsg.2007.09.002. Epub 2007 Dec 4. PMID 18055171
- [Background] Wang BR, Rowe VL, Ham SW, Han S, Patel K, Weaver FA, Woo K. A prospective clinical evaluation of the effects of intraoperative systemic anticoagulation in patients undergoing arteriovenous fistula surgery. Am Surg. 2010 Oct;76(10):1112-4. doi: 10.1177/000313481007601020. PMID 21105622